CLINICAL TRIAL: NCT00484237
Title: A Randomized, Double-Blind, Multicenter, Parallel Study Evaluating the Safety and Efficacy of Etanercept 10 mg Twice Weekly and 25 mg Once Weekly in Japanese Subjects With Active Rheumatoid Arthritis
Brief Title: A Study Evaluating 10 mg and 25 mg Doses of Etanercept in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A1-3324
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

INTERVENTIONS:
Drug: etanercept

SUMMARY:
This study will compare the safety and efficacy for two regimens of etanercept in patients with rheumatoid arthritis (RA). The two regimens to be compared are a 25mg twice weekly regimen and a 50mg once weekly regimen.

DETAILED DESCRIPTION:
This study will compare the safety and efficacy for two regimens of etanercept in patients with rheumatoid arthritis (RA). The two regimens to be compared are a 25mg twice weekly regimen and a 50mg once weekly regimen.

ELIGIBILITY:
Inclusion Criteria:

* Presence of >6 swollen joints and >6 tender joints
* Inadequate response to at least one disease modifying anti-rheumatic drug (DMARD)
* Have not been treated with a DMARD for at least 4 weeks prior to the baseline visit

Exclusion Criteria:

* Previous treatment with etanercept, antibody to TNFα, or other TNFα inhibitors
* Received investigational drugs within 6 months of the baseline visit
* Received intra-articular hyaluronic acid injections within 4 weeks of the baseline visit

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary comparison of the study will be the change of DAS28-4ESR scores from baseline (week 0) between the 10 mg BIW group (at week 12) and the 25 mg QW group (at week 12).

SECONDARY OUTCOMES:
ACR 20, 50, and 70; Number of swollen joints (68 joints); Number of painful joints on pressure or motion (71 joints); Physician global assessment; Patient global assessment; Duration of morning stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (13):
- Japan (13):
  - Goshogawara, Aomori
  - Choseigun, Chiba
  - Yotsukaidō, Chiba
  - Fukuoka, Fukuoka
  - Fukushima, Fukushima
  - Higashihiroshima, Hiroshima
  - Katoh, Hyōgo
  - Sagamihara, Kanagawa
  - Kumamoto, Kumamoto
  - Sendai, Miyagi
  - Nagano, Nagano
  - Sasebo, Nagasaki
  - Ōita, Oita Prefecture